CLINICAL TRIAL: NCT07270224
Title: Motor Imagery Ability, Hand Mental Rotation and Performance Outcomes in Female Volleyball Players: A Comparative Cross-sectional Study
Brief Title: Motor Imagery, Hand Mental Rotation, and Performance in Female Volleyball Players
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ayse Yazgan, Principal Investigator, Medipol University
Other Study IDs: MedipolU-OP-AY-03
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Motor Imagery; Volleyball; Reaction Time; Vertical Jump Performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female Volleyball Players: Female athletes currently participating in competitive volleyball; no intervention applied.
- Controls Group: Female individuals not engaged in regular physical activity; no intervention applied.

SUMMARY:
This comparative cross-sectional study investigates the relationship between motor imagery (MI) ability, hand mental rotation (HMR), and performance outcomes in female volleyball players. Volleyball is a high-speed, cognitively demanding sport requiring precise motor coordination, rapid decision-making, and explosive movements. MI-the mental simulation of movement-and HMR-the cognitive manipulation of hand orientation-are critical for motor planning and execution. The study has two primary objectives: (1) to compare MI ability and HMR performance between female volleyball players and sedentary controls, and (2) to evaluate associations between MI/HMR scores and reaction time as well as vertical jump performance among volleyball players. The investigators hypothesize that volleyball players will exhibit superior MI and HMR abilities compared to controls, and that higher MI and HMR scores will correlate with faster reaction times and greater vertical jump height. Findings from this study will elucidate the cognitive-motor mechanisms underlying athletic performance and may inform training strategies to enhance neuromotor efficiency in sport-specific contexts.

ELIGIBILITY:
Inclusion Criteria: Volleyball Group

* Female participants aged 18-25 years
* Licensed professional volleyball players competing in national or regional leagues
* Currently playing an official main or secondary position
* Minimum of 5 years of professional volleyball experience
* Actively competing in volleyball for at least 1 year
* Training more than 10 hours per week
* No injury in the past 6 months that prevented participation in training or matches
* Ability and willingness to participate voluntarily
* Provided written informed consent

Inclusion Criteria: Control Group

* Female participants aged 18-25 years
* No history of participation in professional or recreational overhead sports
* No lower extremity injury within the past 6 months
* Less than 1 hour per week of structured exercise within the past 6 months
* No previous licensed sports participation
* Provided written informed consent

Exclusion Criteria (Applied to Both Groups)

* Neurological, orthopedic, or systemic diseases
* History of lower extremity injury in the past 6 months
* Any pain, pathology, or instability affecting the upper or lower extremities
* Regular medication use
* Visual or hearing impairments
* Diagnosed cognitive or attention disorders

Ages: 18 Years to 25 Years | Sex: Female
Age Groups: Adult
Study Population: The study population consists of licensed female volleyball players competing in regional leagues and healthy female adults with no history of professional sports participation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2025-11-10 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Mental Chronometry Test | Baseline (single assessment during the initial study visit)
  Mental chronometry ratio calculated as |Actual Time - Imagined Time| / Actual Time, measured during five actual vertical jumps and five imagined vertical jumps. Lower values indicate better motor imagery performance. Time measured in seconds using a stopwatch; ratio is unitless.

SECONDARY OUTCOMES:
Hand Mental Rotation Task | Baseline
  Mean response time (milliseconds) for left/right hand discrimination tasks in the Orientate® application. Lower values indicate faster cognitive processing related to mental rotation.
Reaction Time (ms) | Baseline
  Mean reaction time across three trials measured using the BlazePod® wireless LED sensor system. Participants respond to visual stimuli with their dominant hand. Lower values indicate better reaction performance.
Vertical Jump Height (cm) | Baseline
  Mean jump height calculated from three countermovement jumps recorded and analyzed using the My Jump 2 smartphone application. Higher values indicate better lower-limb explosive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Yazgan, Principal Investigator — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University, Istanbul, Beykoz
  - Ayşe Yazgan, Bakırköy, Istanbul